CLINICAL TRIAL: NCT05747456
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study of IPN-21-SENSE, a Novel Hyaluronic Acid Based Gel for Volume Deficiency in the Mid-face
Brief Title: Study of a Novel Hyaluronic Acid Based Gel for Volume Deficiency in the Mid-face (FaceHyal)
Acronym: FaceHyal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIV-IPN-21-SENSE-01
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Volume Deficiency in the Mid-Face; Aging; Aesthetics
Keywords: Mid-Face; Hyaluronic Acid; Volume; Aging; Aesthetics

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, No-Treatment Controlled Trial. Subjects will be randomized (5:1 ratio) to the IPN-21-SENSE (treatment) arm or the no-treatment control arm.
  After 24 weeks, the no-treatment control arm (delayed treatment group) will receive their first treatment and will then follow the same schedule as the initial treatment group. After the no-treatment control group receives treatment, data from both groups will be pooled.
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint is assessed through objective measures of facial volume, obtained using standardized, three-dimensional (3D), digital photographic images. Measurement will be made by an independent expert who will be blinded, as image files will not reveal subject treatment randomization, or the time point at which the image was taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPN-21-SENSE Treatment Group (Experimental): Subjects randomized (5:1 ratio) to receive an initial treatment with IPN-21-SENSE Crosslinked Hyaluronic Acid Gel up to 8mL, based on the PI's assessment, in combination with the aesthetic goal of the subject, then an optional touch-up treatment session 4 weeks later, up to 4mL.
  Interventions: Device: IPN-21-SENSE
- No-Treatment Control Group, then Delayed Treatment with IPN-21-SENSE (Other): No-Treatment for the first 6-month, then subjects will receive a delayed treatment with IPN-21-SENSE Crosslinked Hyaluronic Acid Gel up to 8mL, based on the PI's assessment, in combination with the aesthetic goal of the subject, then an optional touch-up treatment session 4 weeks later, up to 4mL.
  Interventions: Device: IPN-21-SENSE

INTERVENTIONS:
Device: IPN-21-SENSE — Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek at the first session, on each side of the face.
  Up to 1.0 mL in the zygomaticomalar region and optionally up to 1.0 mL in the anteromedial cheek for the optional touch-up session, on each side of the face.
  Arms: IPN-21-SENSE Treatment Group
Device: IPN-21-SENSE — Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek at the first session, on each side of the face.
  Up to 1.0 mL in the zygomaticomalar region and optionally up to 1.0 mL in the anteromedial cheek for the optional touch-up session, on each side of the face.
  Arms: No-Treatment Control Group, then Delayed Treatment with IPN-21-SENSE

SUMMARY:
The primary objective of the study is to demonstrate the superiority of IPN-21-SENSE versus no treatment at 24 weeks after baseline for the creation or restoration of volume deficit in the mid-face.

DETAILED DESCRIPTION:
This is a prospective, randomized, no-treatment controlled clinical trial of a proposed class III medical device. This study is designed to demonstrate clinical safety and performance of the IPN-21-SENSE dermal filler in the restoration or creation of volume in the mid-face.

The objective of this study is to demonstrate the superiority of IPN-21-SENSE versus no treatment at 24 weeks after baseline for the creation or restoration of volume deficit in the mid-face.

Assessment of superiority will be based on 3D analysis of the volumetric change, using a validated imaging system.

Effectiveness of IPN-21-SENSE will be demonstrated if the mean volumetric change at 24 weeks after baseline from pre-treatment in the treatment group is statistically superior to the mean change in the delayed treatment (control) group.

In total, approximately 90 subjects will be enrolled across two study centers in France and Poland.

Subjects will be randomized to the treatment group or delayed treatment (control) group at a 5:1 ratio (i.e., there will be 5 more subjects treated with IPN-21-SENSE at baseline as compared to subjects who will be in the no-treatment (control) group and who will receive a delayed treatment with IPN-21-SENSE at 24 weeks after baseline).

The total duration of subject participation ranges from 18 months (treatment group) to 24 months (delayed treatment (control) group). Overall study duration including the enrolment period is expected to take approximately 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 84 years.
* Seeking correction of the mid-face volume deficit, and agrees with the recommendation of the Investigator.
* Accept the obligation not to receive any other facial procedures or treatments impacting facial volume augmentation at any time during the study.
* Able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
* Psychologically able to understand the study related information and to give a written informed consent
* Have voluntarily provided written informed consent to participate in the study, and use of data privacy (sign the ethics committee approved Informed Consent Form), prior to any study-related procedure being performed.
* Female of childbearing potential (sexually active, not sterile, nor postmenopausal for at least 1 year) must have a negative urine pregnancy test (UPT) at Visit 1 (or Visit 1b), and use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and for the duration of the study.
* Affiliated to a health social security system.

Exclusion Criteria:

In terms of population:

* Pregnant or breastfeeding woman, or planning a pregnancy during the study.
* Scars, moles, tattoo, or anything on the Mid-face which might interfere with the evaluation.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or who is in an exclusion period of one.
* Subject having received 4,500 Euros in indemnities for participation in research involving human beings in France in the past 12 months, including participation in the present study (for France only).

In terms of associated pathology:

* Subject presenting any symptom which can be related to a medical condition that is likely to make the subject not being compliant with the study schedule, at the discretion of the investigator.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject suffering from active inflammatory and/or infectious cutaneous disorders in or near the studied zones (e.g., herpes, acne). Subject with recurrent herpes in the Midface area is eligible if asymptomatic at time of inclusion.
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
* Subject with any history of healing disorders.
* Subject having history of allergy or anaphylactic shock including hypersensitivity to hyaluronic acid, to lidocaine, or to antiseptic solution or any other amide type local anaesthetics.
* Subject presenting a history of severe, evolutive, unstable, or recent allergies.
* Subject suffering from porphyria.
* Subject with a cancer in areas close to the injection site, and subjects with a melanoma
* Subject with epilepsy or severe respiratory or cardiac function disorder.
* Subject with severe renal or hepatic functions disorders.

Relating to previous or ongoing treatment:

* Subject having received treatment with a laser or ultrasound, a dermabrasion, a surgery, a deep chemical peeling, or other ablative procedure on the midface area within the past 12 months prior to inclusion.
* Subject having received injection with a resorbable filling product in the midface area, defined as the zygomaticomalar and the anteromedial cheek regions, within the past 18 months prior to inclusion.
* Subject having received injection with a resorbable filling product in the nasolabial folds and/or the eye shadows, within the past 12 months prior to inclusion.
* Subject having received injection with a resorbable filling product in any part of the body of more than 8 mL within the past 12 months prior to inclusion.
* Subject having received at any time injection with a slowly resorbable filling product (e.g., polylactic acid, calcium hydroxyapatite, combinations of ha and hypromellose) or with a non-resorbable filling product (e.g. polyacrylamide or silicone).
* Subject having received at any time a treatment with tensor threads in the Midface area, or a surgery in the mid-face, or who plan to undergo any of these procedures during the study.
* Subject under medications which may cause lipo-atrophy.
* Subject using medication that reduce or inhibit hepatic metabolism (cimetidine, beta-blockers, etc)
* Subject being under immunosuppressive therapy.
* Subject undergoing a topical treatment on the test area or a systemic treatment:
* Antihistamines during the 3 days prior to study start
* Immunosuppressors and/or corticoids during the 4 weeks prior to study start
* Retinoids during the 6 months prior to study start.
* Subject having received a covid vaccine less than 4 weeks before the IPN-21-SENSE injection

Ages: 30 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Mid-Face Volumetric change | 24 weeks after baseline
  Mean volumetric change between the treatment group and no-treatment control group at 24 (V4) weeks after baseline (V1)

SECONDARY OUTCOMES:
Mid-Face Volumetric change | 4, and 12 weeks after baseline
  Mean volumetric change between the treatment group and no-treatment control group at 4 (V2) and 12 (V3) weeks after baseline (V1)
Mid-Face Volumetric change | 4, 12, 24, 48, and 72 weeks after initial treatment
  Mean volumetric change between pre-treatment and directly after treatment at V1 (or V1b), and 4 (V2/V2b), 12 (V3/V3b), 48 (V5), and 72 (V6) weeks after initial treatment, in both groups pooled.
Global Aesthetic Improvement, by the Subjects | 4, 12, and 24 weeks after baseline
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Subjects, between the treatment group and no-treatment control group.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Subjects | 4, 12, 24, 48, and 72 weeks after initial treatment
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Subjects, in both groups pooled.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Investigators | 4, 12, and 24 weeks after baseline
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Investigators, between the treatment group and no-treatment control group.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Investigators | 4, 12, 24, 48, and 72 weeks after initial treatment
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Investigators, in both groups pooled.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
FACE-Q, by the Subjects | Baseline, and 4, 12, and 24 weeks after baseline
  Rash-transformed score of the FACE-Q, assessed by the Subjects, between the treatment group and no-treatment control group.
  FACE-Q is a patient-reported outcome (PRO) measure that can be used to measure outcomes of aesthetic facial procedures and products from the patient's perspective, composed of a set of independently functioning scales/checklists. In this study; two scales are assessed:
  1. FACE-Q - Satisfaction with cheekbones: This questionnaire consists of 10 items, and measures the appearance of cheekbones with items that ask about shape, contour and symmetry, as well as how attractive, high and well-defined the cheekbones look.
  2. FACE-Q - Satisfaction with outcome. This questionnaire consists of 6 items, and measures satisfaction with the result of a facial procedure, e.g., pleased with the result, result is fantastic.
  The total score is converted to a score from 0 to 100, with higher scores reflect a better outcome.
FACE-Q, by the Subjects | Initial treatment, and 4, 12, 24, 48, and 72 weeks after initial treatment
  Rash-transformed score of the FACE-Q, assessed by the Subjects, in both groups pooled.
  FACE-Q is a patient-reported outcome (PRO) measure that can be used to measure outcomes of aesthetic facial procedures and products from the patient's perspective, composed of a set of independently functioning scales/checklists. In this study; two scales are assessed:
  1. FACE-Q - Satisfaction with cheekbones: This questionnaire consists of 10 items, and measures the appearance of cheekbones with items that ask about shape, contour and symmetry, as well as how attractive, high and well-defined the cheekbones look.
  2. FACE-Q - Satisfaction with outcome. This questionnaire consists of 6 items, and measures satisfaction with the result of a facial procedure, e.g., pleased with the result, result is fantastic.
  The total score is converted to a score from 0 to 100, with higher scores reflect a better outcome.
Wrinkle Severity Rating Scale (WSRS), by the Investigators. | 4, 12, and 24 weeks after baseline
  Nasolabial Fold Severity using the wrinkle severity rating scale (WSRS), assessed by the Investigators, between the treatment group and no-treatment control group.
  The WSRS (Wrinkle Severity Rating Scale) is a 5-point rating scale to determine the severity of the nasolabial folds (NLF), with lower scores mean better condition (less severity), with 1 means "Absent - No visible NLF, continuous skin line" and 5 means "Extreme - Extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched".
Wrinkle Severity Rating Scale (WSRS), by the Investigators. | 4, 12, 24, 48, and 72 weeks after initial treatment
  Nasolabial Fold Severity using the wrinkle severity rating scale (WSRS), assessed by the Investigators, in both groups pooled.
  The WSRS (Wrinkle Severity Rating Scale) is a 5-point rating scale to determine the severity of the nasolabial folds (NLF), with lower scores mean better condition (less severity), with 1 means "Absent - No visible NLF, continuous skin line" and 5 means "Extreme - Extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched".
Ease of sculpting and massaging, by the Investigators | Initial treatment, and 4 weeks after initial treatment
  Ease of sculpting and massaging of the HA gel, assessed by the investigator after each treatment session, on a 5-point scale ranging from "Very easy" to "Very difficult", in both groups pooled.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia MOREL-MANDRINO, MD, Principal Investigator — Eurofins Dermscan, Villeurbanne, FRANCE
Locations (1):
- Eurofins Dermscan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No